CLINICAL TRIAL: NCT06154954
Title: The Value of Composite Measurements of Extracellular Matrix Protein1, Testis-Expressed Gene 101, and Lectin Galactoside-binding Protein in Predicting Surgical Sperm Retrieval in Men With Non-Obstructive Azoospermia
Brief Title: Testicular Proteins for Sperm Retrieval Prediction Protein1, Testis-Expressed Gene 101, and Lectin Galactoside-binding Protein in Predicting Surgical Sperm Retrieval in Men With Non-Obstructive Azoospermia
Acronym: Genomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Wael Ragab, Lecturer, Cairo University
Other Study IDs: MD-2024
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Non-obstructive Azoospermia
MeSH Terms: interventions — Semen Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Semen analysis — Semen analysis for extracellular matrix proteins analysis

SUMMARY:
Generally, azoospermia is characterized as obstructive (OA) or nonobstructive (NOA). Surgical spermatozoa retrieval results vary in success rates. Proposing Intracytoplasmic Sperm Injection (ICSI) to infertile couples with NOA depends on spermatogenesis, testicular histology, and the ability to extract live spermatozoa from testis biopsy pieces.

Unfortunately, only 50% of testicular sperm extraction (TESE) results are positive (Zarezadeh et al., 2021). Repeating sperm retrieval can cause TESE-induced hypoganadism, including reduced testicular volume, erectile dysfunction, and testosterone deficiency (Eliveld et al., 2018; Okada et al., 2002; Ozturk et al., 2011; Altinkilic et al., 2017; Akbal et al., 2017; Binsaleh et al., 2017). The prognostic efficacy of hormonal, molecular, cytological, and biochemical indicators for effective sperm recovery is limited (Corona et al., 2019). Molecular, biochemical, clinical, and histopathological characteristics that identify NOA males with advanced spermatogenesis foci up to the spermatozoon stage are crucial for therapeutic purposes.

Recent research suggests that seminal protein expression patterns change dramatically between azoospermic and fertile males (Zhang et al., 2021). TEX101 is a membrane protein only produced by testicular germ cells and shed into seminal plasma (SP). Research suggests that Tex101 malfunctions may impact male fertility (Jarvi et al., 2021). TEX101 is a germ cell mono-specific marker present on sperm, round spermatids, and spermatocytes. At a threshold of >5 ng/mL, TEX101 can distinguish NOA with Sertoli-cell only syndrome from other testis histologies, such as hypospermatogenesis (67% specificity, 100% sensitivity) or maturation arrest (54% sensitivity, 100% specificity) (Drabovich et al., 2013). ECM1, an epididymal mono-specific marker, was below detection limits in males with OA semen but present in detectable levels.

Research Template 3: Final Version: April 2019 NOA amounts in males. Clinical immunoassays of ECM1 and TEX101 can predict sperm retrieval outcomes for assisted reproduction and lower the cost of diagnosing azoospermia.

ELISA confirms that the lectin galactoside-binding, soluble 3 binding protein (LGALS3BP) is expressed throughout the male genital tract. Its physiological role in cell-to-cell interaction through extracellular matrix suggests a possible role in spermatogenesis, particularly in the late stage, despite not being a germ-cell specific marker (Cannarella et al., 2020). Patients with a good result of TESE had significantly greater levels of LGALS3BP in the SP. A cut-off of 153 ng/mL was observed with 100% sensitivity and 45% specificity. Freour et al. (2013) identified a key issue in their analysis due to the small number of instances (n=40) with lower AUC values. Araujo and Bertolla (2021) propose that LGALS3BP may predict TESE success in NOA patients before ICSI.

DETAILED DESCRIPTION:
Azoospermia is mainly classified as obstructive azoospermia (OA) or nonobstructive azoospermia (NOA). Surgical retrieval of spermatozoa yields various success rates. The chance for proposing Intracytoplasmic Sperm Injection (ICSI) to infertile couple in case of NOA depends on spermatogenesis, testicular histology and on the possibility to retrieve live spermatozoa from testis biopsy fragments.

Unfortunately, this favorable outcome is obtained in only 50% of testicular sperm extraction (TESE) (Zarezadeh et al., 2021). Repeating the sperm retrieval procedure may lead to TESE induced hypoganadism (Eliveld et al., 2018) including the chance of reduced testicular volume (Okada et al., 2002, Ozturk et al., 2011, Altinkilic et al., 2017), the probability of erectile dysfunction (Akbal et al., 2017) and testosterone deficiency (Altinkilic et al., 2017, Binsaleh et al., 2017). Various hormonal, molecular, cytological, biochemical predictive parameters for successful sperm recovery offer limited predictive power (Corona et al., 2019). It is obvious that the establishment of molecular, biochemical, clinical or histopathological parameters that have a role in identifying subpopulations of NOA men positive for foci of advanced spermatogenesis, up to the spermatozoon stage, has great clinical importance. Recent studies demonstrated that the seminal protein expression pattern could differ significantly between azoospermic patients and fertile men (Zhang et al., 2021). Testis-expressed gene 101 (TEX101) is a cell membrane protein exclusively expressed by testicular germ cells and shed into seminal plasma (SP). There have been indications that the malfunction of Tex101 may affect male fertility (Jarvi et al., 2021). TEX101 is a germ cell mono-specific marker found on sperm, round spermatids, and spermatocytes. TEX101, at a threshold >5 ng/mL, could differentiate NOA underlined by Sertoli-cell only syndrome from NOA due to other testis histology (e.g., hypospermatogenesis, with a 67% specificity and a 100% sensitivity, or maturation arrest, with a 54% sensitivity and a 100% specificity) (Drabovich et al., 2013). ECM1 is an epididymal mono-specific marker which was below detection limits for men with OA, but present in the semen in detectable Research Template 3 Final Version: Ap ril 2019 amounts in men with NOA. Clinical immunoassays of extracellular matrix protein1 (ECM1) and TEX101 have the potential to facilitate prediction of the outcome of sperm retrieval procedures used for assisted reproduction, and reduce the total cost of azoospermia diagnosis. The lectin galactoside-binding, soluble 3 binding protein (LGALS3BP) is expressed in the whole male genital tract, with an expression level compatible with ELISA confirmation method, and because its physiological role in cell to cell interaction through extracellular matrix supports a possible role in spermatogenesis especially the late stage of spermatogenic activity, even if it is not a germ-cell specific marker (Cannarella et al., 2020). Significantly higher levels of lectingalactoside-binding, soluble 3 binding protein (LGALS3BP) in the SP were found in patients with a positive outcome of TESE. The cut-off of 153 ng/mL was reported with a sensitivity of 100% and a specificity of 45%. However, the limited number of cases (n=40) with a consequent lower AUC value represent a major flaw in that study (Freour et al., 2013). Araujo and Bertolla suggest that LGALS3BP could potentially be used as a predictive marker of success of TESE in NOA patients before ICSI (Araujo and Bertolla 2021).

ELIGIBILITY:
Inclusion Criteria:

* Men with Non-obstructive azoospermia

Exclusion Criteria:

1. Sex reversal syndrome.
2. Macro-deletion on the Y chromosome (To those accepting the chromosomal study)
3. AZF a, AZF b microdeletion (To those accepting the Y chromosome microdeletion analysis).
4. Obstructive azoospermia.
5. Undescended testis.
6. Hypogonadotrophic Hypogonadism
7. Testicular procedures and operations -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males 46,XY
Study Population: Azoospermic patients whom are scheduled for TESE operation attending at Andrology clinic, Kasr Al Ainy hospital.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Calculating the cut off level of the following markers a. ECM, b. TEX 101 and c. LAGALS3BP | 6 months
  These proteins if present, they would provide the highest yield of sperms

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University hospital, department of andrology, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No